CLINICAL TRIAL: NCT02069301
Title: Development of an Integrated Microfinance and Depression Care Program for Women
Brief Title: Evaluation of an Integrated Microfinance and Depression Care Program for Women
Acronym: LIFE-DM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Danang Psychiatric Hospital (Other)
Responsible Party: Principal Investigator, Victoria K. Ngo, PhD, Behavior Scientist, RAND
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5R34MH094648-02 (NIH); 5R34MH094648-02 (NIH)
Record Dates: First submitted 2014-02-10; First posted 2014-02-24 (Estimated); Last update posted 2017-11-30 (Actual); Status verified 2017-11

CONDITIONS: Depression
Keywords: Behavior Activation; Problem solving therapy; Depression Treatment; depression care integration; microfinance; livelihood
MeSH Terms: conditions — Depression | interventions — Therapeutics; Fluoxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Integrated Depression/Microfinance Group (Experimental): LIFE-DM is a Depression and Microfinance integrated program using behavior activation and problem solving therapy applied to both depression and livelihood. Livelihood support include microfinance loans, personal finance, and income-generation skills.
  Interventions: Behavioral: Integrated Depression/Microfinance Group; Other: Treatment as Usual; Other: Livelihood Support
- Treatment as Usual (Other): Currently treatment as usual in this province includes national guidelines for antidepressant care for depression and referral for microfinance/livelihood programs
  Interventions: Other: Treatment as Usual

INTERVENTIONS:
Behavioral: Integrated Depression/Microfinance Group — LIFE-DM Integrated Depression and Microfinance group, uses behavior activation and problem solving therapy skills to teach patients how to manage mood and reach livelihood goals.
  Other Names: LIFE-DM Group
  Arms: Integrated Depression/Microfinance Group
Other: Treatment as Usual — National Guideline for antidepressant care
  Other Names: Guideline antidepressant care; Fluoxetine, Amitrytaline; other antidepressants
Other: Livelihood Support — Livelihood support, including group-based loans to develop small enterprise, personal finance management education, business management skills, vocational training, and rotating-credit savings program.
  Other Names: Microfinance loans
  Arms: Integrated Depression/Microfinance Group

SUMMARY:
The study evaluates LIFE-DM, an integrated microfinance and collaborative care intervention by comparing it to enhanced treatment as usual (national guideline antidepressant care and referral to microfinance resources) in Vietnam. Intervention effects at baseline, 6 month, and 12 month follow-up on patient outcomes, including depression, anxiety, quality of life, functioning, self-efficacy, satisfaction, and income will be compared across the two conditions.

DETAILED DESCRIPTION:
Depression is one of the largest contributors to the world's health burden. Prior work in the Partners in Care study has shown that evidence-based service delivery programs for depression can improve health outcomes in depressed patients, and especially in minorities, largely overcoming disparities in outcomes from care between whites and minorities. Effective treatments exist, but they do not reach many depressed individuals, especially in resource-poor communities--ethnic minorities, rural residents in the United States, and individuals in most of the developing world.

Women, in particular, are at risk for depression and poverty. Integrating programs that treat depression and address livelihood concerns may improve engagement in depression treatment and improve mental health and functioning for patients in low-resource settings. The proposed study would integrate depression care with existing "microfinance" programs, which provide poverty-alleviation services including small loans, savings programs, and vocational training to women.

This project will (1) conduct qualitative studies of barriers and facilitators of women's successful use of existing depression care and microfinance programs; (2) adapt and integrate the depression care and microfinance services; (3) train Women's Union facilitators to deliver the integrated depression care and microfinance program; and conduct evaluation of LIFE-DM program to assess acceptability, feasibility, and preliminary effectiveness. The non-randomized control trial compares the integrated microfinance and collaborative care intervention with enhanced treatment as usual (national guideline antidepressant care and referral to microfinance resources) at the Women's Union in Danang city in Vietnam.

ELIGIBILITY:
Inclusion Criteria:

* depression, low-income

Exclusion Criteria:

* psychosis, mania, substance abuse, high suicide risk, physical disabilities, significant cognitive impairments

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 166 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Change in Depression Score from the Patient Health Questionnaire | 0, 6, 12 months
  The PHQ-9 is a nine-item validated tool measuring depressive symptoms based on DSM-IV criteria. The answers are rated on a scale from zero (not at all) to three (nearly every day). Total scores range from 0-27, subdivided into five categories of depression severity: 1 to 4 is minimal; 5 to 9 is mild; 10 to 14 is moderate; 15 to 19 is moderate-severe; and 20 and above is severe. The PHQ-9 has been widely used internationally including in Vietnam.

SECONDARY OUTCOMES:
Change in Quality of Life Score from Quality of Life and Enjoyment and Satisfaction Questionnaire | 0, 6, 12 months
  The Quality of Life Enjoyment and Satisfaction Questionnaire is a self-report measure designed to enable investigators to easily obtain sensitive measures of the degree of enjoyment and satisfaction experienced by subjects in various areas of daily functioning. The summary scores were found to be reliable and valid measures of these dimensions in a group of depressed outpatients. The Q-LES-Q measures were related to, but not redundant with, measures of overall severity of illness or severity of depression within this sample. These findings suggest that the Q-LES-Q measures may be sensitive to important differences among depressed patients that are not detected by the measures usually employed.
Change in Self-Efficacy Score from Self Efficacy Survey | 0, 6, 12 months
  Items were developed to assess effectiveness of a goal-setting and planning intervention (Macleod et al., 2008). Self-efficacy is assessed via 4-items that measure locus of control, materials and skills to complete goals, confidence, and optimism. Self-efficacy is rated on a 9-point scale from 1 ("Not at all") to 9 ("To a great extent").
Change in Social Support Index from Medical Outcome Study Social Support Survey | 0, 6, 12 months
  A brief, multidimensional, selfadministered, social support survey that was developed for patients in the Medical Outcomes Study (MOS), a two-year study of patients with chronic conditions. This survey was designed to be comprehensive in terms of recent thinking about the various dimensions of social support.
Change in health and mental health functioning scores from Medical Outcomes Study Short Form Health Survey (SF-12) | 0, 6, 12 months
  The SF-12v2 is a 12-item survey that measures the same eight domains of health. The domains scores are summarized into two composite scores: Physical Component Summary and Mental Component Summary scores. The survey is a brief, reliable measure of overall health status. It is useful in large population health surveys and has been used in Vietnamese populations.
Change in Anxiety Symptom Score from Generalized Anxiety Disorder (GAD-7) Scale | 0, 6, 12 months
  The GAD-7 is a 7-item anxiety scale used for screening and assessing symptom severity of GAD. GAD and depression symptoms frequently occurred together, but factor analysis confirmed them as distinct dimensions, and they had independent effects on functional impairment and disability. Self-report and interviewer-administered versions of GAD-7 were in good agreement.
Change in Behavior Activation Score from the Behavior Activation for Depression Scale Short Form (BADS-SF) | 0, 6, 12 months
  The abbreviated BADS-SF is a nine-item scale measuring factors expected to change as a function of behavioral activation, including activation and avoidance
Change in household wealth indicators from Economic Well-Being Inventory | 0, 6, 12 months
  The economic well-being inventory collect various indicators of self-reported household wealth: housing materials, land ownership, home ownership, and selling and purchasing of assets such as livestock and durable goods (car, bicycle, radio, TV), as well as income, savings, and debt. This economic well-being inventory was used in the Danang Household Mental Health Survey.
Change in number and type of income generating activities from the Employment and business Activities Questionnaire | 0, 6, 12 months
  We developed questionnaire to measure income generating activities, which include questions about participation and number of hours in types of employment and income generating activities in Low-Income countries, including formal salaried employment, farming and planting food, selling goods and services, property rentals, etc.
Treatment Acceptability Score from Help-Seeking Behavior Questionnaire | 0, 6, 12 months
  This measure consists of items that assesses 1) resources in the community, 2) participant's help seeking history, 3) perceived effectiveness, and 4) acceptability of a variety of strategies used for depression care.
Depression Stigma Score from the Depression Stigma Questionnaire | 0, 6, 12 months
  18 item questionnaire about perceived and personal stigma related to depression.
Social Capital Score from Social Capital Assessment Tool | 0, 6, 12 months
  The short version of the Adapted Social Capital Assessment Tool (SASCAT) is a nine-item tool measures the structural (quantity of social relationships) and cognitive (quality of social relationships) components of social capital as well as citizenship. The measure derived from the Adapted Social Capital Assessment Tool (A-SCAT) (Harpham et al., 2002). The measures has been used in many international settings, including developing countries.
Total Score Client Service Satisfaction Questionnaire | 0, 6, 12 months
  A standardized measure with strong psychometric properties that could be used to assess general satisfaction across varied health and human services. The CSQ Scales® (CSQ) measure may be used to assess client satisfaction with mental health services, as a program evaluation tool, or to assess client satisfaction within and across programs (intra- or inter-program) and demographic groups.
Number of Participants Demonstrating Mental Health Literacy with Depression Vignette | 0, 12 months
  Vignette describes someone with the minimal number of symptoms necessary for major depression (according to DSM description). Respondents were asked an open-ended question, ''What would you say, if anything, is wrong with Mary?'' Only answers including " depression " are considered a correct response.
Number of Participants with Depression Diagnosis - MINI International Neuropsychiatric Interview, Version 6.0 (MINI) | 0, 6, 12 months
  The MINI is a brief structured psychiatric interview used to diagnose for multiple axis I DSM-IV mental disorders. In this study, the MINI is used to assess for major depressive episodes. Using DSM-IV criteria (at least 5 symptoms of depression over a 2 week period; endorsement of depressed mood or anhedonia were necessary for diagnosis) the interviewers can distinguish between past, current, and recurrent episodes of depression. The MINI is a reliable and valid alternative to the longer Structured Clinical Interview for Diagnostic. The MINI has been used widely in developing countries and administered by non-mental health providers.

CONTACTS AND LOCATIONS:
Overall Officials: Victoria K Ngo, PhD, Principal Investigator — RAND
Locations (4):
- Vietnam (4):
  - Hoa Cuong Bac Commune Health Station, Da Nang
  - Hoa Cuong Nam Commune Health Station, Da Nang
  - Hoa Hiep Nam Commune Health Station, Da Nang
  - Hoa Minh Commune Health Station, Da Nang

REFERENCES:
- [Result] Ngo VK, Weiss B, Lam T, Dang T, Nguyen T, Nguyen MH. The Vietnam Multicomponent Collaborative Care for Depression Program: Development of Depression Care for Low- and Middle-Income Nations. J Cogn Psychother. 2014;28(3):156-167. doi: 10.1891/0889-8391.28.3.156. PMID 25568593